CLINICAL TRIAL: NCT07259863
Title: Clinico_Epidemiological Profile Of Acquired Aplastic Anemia Among Children At Assiut Governorate.
Brief Title: Clinico-Epidemiological Profile Of Acquired Aplastic Anemia Among Children At Assiut Governorate .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Ramadan Hassanein Hassan, Assistant Lecturer, Assiut University
Other Study IDs: Aplastic anemia in children .
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Acquired Aplastic Anaemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational case series study no intervention — Assessment the clinical presentation and epidemiological profile of children with acquired aplastic anemia. 2.Determining the possible risk factors and associated conditions contributing to the development of acquired aplastic anemia.

SUMMARY:
1. Assessment the clinical presentation and epidemiological profile of children with acquired aplastic anemia.
2. Determining the possible risk factors and associated conditions contributing to the development of acquired aplastic anemia.

DETAILED DESCRIPTION:
Aplastic anaemia is a term describing the common findings of pancytopenia and marrow hypoplasia from arising variety of disease states, including acquired aplastic anaemia and a variety of congenital marrow failure states(1). The global incidence of paediatric AA varies geographically, with rates of 2 to 3 cases per million per year in Europe, but higher in East Asia and certain developing regions(2) .Among Egyptian Children, inherited bone marrow failure syndromes (BMFS), including AA, constitute about 10-15%of all BMFS and up to 30% of paediatric BMFS ,with an average of 65 cases per million live births each year .Acquired AA remains the predominant from in older children and adolescent , while inherited forms are more common in younger children(3).The clinical presentation of aplastic anaemia regularly consists of symptoms associated with pancytopenia, including fatigue, pallor, bruising, bleeding, and extended susceptibility to infections(4). Identified etiologic risk factors include infections of viral origin, such as hepatitis-associated, Epstein-Barr, parvovirus, human immunodeficiency virus, varicella zoster, measles and other viruses, as well as exposure to toxic chemicals (e.g. benzene, pesticides and insecticides) and ionizing radiation (5). Over the last three decades, bone marrow transplantation (BMT) from a matched related donor (MRD) has been the treatment of choice for children with acquired AA (6) The Rationale of our study: aplastic anaemia in children is a serious ,life threatening bone marrow failure syndrome ,often resulting from immune-mediated destruction of hematopoietic stem cell triggered by factors such as viral infections, environmental toxin, or genetic predispositions and requires precise diagnosis to distinguish from inherited bone marrow failure syndromes or hypoplastic myelodysplastic syndrome to guide appropriate treatment strategies .

The Research question: What is the clinico-epidemiological profile of acquired aplastic anaemia among children at Assiut governorate.

ELIGIBILITY:
Inclusion Criteria:

* 1- Children aged 1-18 years old diagnosed with acquired aplastic anemia 2-Fulfillment of the diagnostic criteria for acquired AA 3-patient with complete medical records,including diagnostic ,labaratory and treatement data 4-Diagnosed or treated at assuit university children hospital and the central health insurance clinic at assuit Governorate (october 2020 to october 2026)

Exclusion Criteria:

* 1-children with congental bone marrow failure syndrome 2-patient with a history of chemotherapy or radiotherapy prior to diagnosis 2-cases with incomplete medical or insufficient medical records that prevented confirmination of diagnosis or extraction of essential study data

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children at 1 to 18 years old diagnosed with acquired aplastic anemia at assuit governorate from october 2020 to october 2026
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Acquired Aplastic Anemia among children | from October 2020 to October 2026
  Determine the clinic-epidemiological profile of acquired aplastic anemia among children at assiut governorate
determine the clinico-Epidemiological profile of acquired aplastic anemia among children at assuit governorate | from october 2020 to october 2026
  To descripe and record clinical characteristic ,management,and outcomes of the included cases

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mohamed Embaby, professor of pediatic, Principal Investigator — Departement of Familly medicine Assuit University

IPD SHARING:
Plan to Share IPD: No